CLINICAL TRIAL: NCT07094113
Title: A Phase 1/1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of AMG 410 Alone and in Combination With Other Agents in Participants With KRAS Altered Advanced or Metastatic Solid Tumors
Brief Title: AMG 410 Alone and in Combination With Other Agents in Participants With KRAS Altered Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20240031
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: KRAS Altered Advanced or Metastatic Solid Tumors
Keywords: Non-small cell lung cancer; NSCLC; Colorectal cancer; CRC; Pancreatic ductal adenocarcinoma; PDAC; AMG 410
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — pembrolizumab; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Monotherapy Dose Exploration (Experimental): Participants will receive escalating doses of AMG 410.
  Interventions: Drug: AMG 410
- Part 1: Food Effect Substudy Cohort (Experimental): A food effect substudy will be conducted. During the substudy, participants will receive AMG 410 under fasted and fed conditions.
  Interventions: Drug: AMG 410
- Part 1: China-specific Cohort (Experimental): Participants identified through regionally approved molecular KRAS testing will receive AMG 410.
  Interventions: Drug: AMG 410
- Part 2: Monotherapy Dose Expansion (Experimental): Monotherapy dose expansion of AMG 410 may proceed in KRAS altered tumors in non-small cell lung cancer (NSCLC), colorectal cancer (CRC), pancreatic ductal adenocarcinoma (PDAC), and other KRAS altered tumor types.
  Interventions: Drug: AMG 410
- Part 3a: Combination Therapy Dose Exploration and Dose Expansion (Experimental): Part 3a allows for AMG 410 dose exploration and expansion in combination with pembrolizumab in KRAS altered advanced or metastatic solid tumors.
  Interventions: Drug: AMG 410; Drug: Pembrolizumab
- Part 3b: Combination Therapy Dose Exploration and Dose Expansion (Experimental): Part 3b allows for AMG 410 dose exploration and expansion in combination with panitumumab in advanced or metastatic CRC and/or PDAC.
  Interventions: Drug: AMG 410; Drug: Panitumumab

INTERVENTIONS:
Drug: AMG 410 — Administered as an oral tablet.
Drug: Pembrolizumab — Administered as an intravenous (IV) infusion.
  Arms: Part 3a: Combination Therapy Dose Exploration and Dose Expansion
Drug: Panitumumab — Administered as an IV infusion.
  Arms: Part 3b: Combination Therapy Dose Exploration and Dose Expansion

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of AMG 410 when administered alone or in combination with other agents in participants with advanced or metastatic solid tumors harboring KRAS alterations.

This is a dose-escalation study in which participants will be assigned to multiple dose levels (DLs) of AMG 410, either as monotherapy or in combination with other agents, followed by expansion cohorts. The goal is to determine the Maximum Tolerated Dose (MTD)-the highest dose with acceptable safety and manageable side effects-or the Recommended Phase 2 Dose (RP2D) of AMG 410 in adult participants with KRAS-altered advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, multinational, open-label Phase 1/1b study designed to evaluate the safety, tolerability, PK, PD, and preliminary antitumor activity of AMG 410 in adult participants with advanced or metastatic solid tumors characterized by KRAS alterations.

The study will begin with a dose-escalation phase, during which AMG 410 will be administered orally, either as monotherapy or in combination with other agents. Dose escalation will follow a model-based approach to identify the MTD or RP2D.

Following dose escalation, additional expansion cohorts may be enrolled at selected dose levels to further characterize the safety profile, PK/PD relationships, and preliminary efficacy in specific tumor types or molecular subgroups.

Participants will continue treatment until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-defined discontinuation criteria. The maximum duration of AMG 410 administration in this study is 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (or > legal age within the country if it is older than 18 years).
2. Pathologically documented, locally-advanced or metastatic malignancy with any missense mutation in the KRAS gene or evidence of KRAS amplification using an analytically validated KRASWT amplification assay.
3. Participants must have no standard of care treatment options or have actively refused such therapy.
4. Able to swallow and retain per oral administered study treatment.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Disease measurable as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), as determined by the site investigator.
7. Adequate organ function.
8. Archival (formalin-fixed, paraffin-embedded [FFPE]) tumor tissue or block collected within 5 years before screening must be available. Participants without archived tumor tissue may undergo tumor biopsy before AMG 410 dosing (Day1).

Exclusion Criteria:

1. Untreated symptomatic central nervous system or leptomeningeal metastases.
2. Uncontrolled pleural effusion and/or ascites.
3. History of other malignancy within the past 5 years.
4. Active systemic infection or symptoms that indicate an acute and/or uncontrolled infection requiring IV antibiotics within 7days prior to the first dose of study treatment.
5. History of arterial or venous thrombosis (eg, stroke, transient ischemic attack, pulmonary embolism, or deep vein thrombosis).
6. Live and live-attenuated vaccines are prohibited within 28 days prior to the first dose of study treatment.
7. History of solid organ transplant.
8. Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, hormonal therapy, or investigational agent) within 28 days of first dose of study treatment.
9. Presence or history of any of the following viral infections: HIV, Hepatitis C, Hepatitis B, and active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
10. Toxicities from prior anti-tumor therapy (including radiotherapy) not having improved to at least Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1.
11. Therapeutic or palliative radiation therapy within 2 weeks of first dose of study treatment.
12. Major surgery within 28 days of first dose of study treatment.
13. History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-04-18 (Estimated); Study Completion 2031-04-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to approximately 3 years
  Clinically significant changes in safety assessments (vital signs, electrocardiograms [ECGs], and clinical laboratory tests) are to be reported as adverse events.
Number of Participants with Serious Adverse Events (SAEs) | Up to approximately 3 years
  Clinically significant changes in safety assessments (vital signs, ECGs, and clinical laboratory tests) are to be reported as adverse events.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of AMG 410 | Up to 85 days
Time to Reach Cmax (Tmax) of AMG 410 | Up to 85 days
Area Under the Concentration-time Curve (AUC) Over the Dosing Interval of AMG 410 | Up to 85 days
Confirmed Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to approximately 3 years
Clinical Benefit per RECIST v1.1 | Up to approximately 3 years
Duration of Response (DoR) per RECIST v1.1 | Up to approximately 3 years
Time to Response (TTR) per RECIST v1.1 | Up to approximately 3 years
Progression-free Survival (PFS) per RECIST v1.1 | Up to approximately 3 years
Overall Survival (OS) | Up to approximately 3 years
Food Effect Substudy Cohort: Cmax of AMG 410 in the Fed and/or Fasted State | Up to 24 days
Food Effect Substudy Cohort: Tmax of AMG 410 in the Fed and/or Fasted State | Up to 24 days
Food Effect Substudy Cohort: AUC Over the Dosing Interval of AMG 410 in the Fed and/or Fasted State | Up to 24 days
Change From Baseline in Tumor Phosphorylated Extracellular Signal Regulated Kinase (pERK) | Baseline up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (27):
- United States (9):
  - City of Hope National Medical Center, Duarte, California
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Siteman Cancer Center - Washington University, St Louis, Missouri
  - Duke Cancer Center, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute Oncology Partners, Nashville, Tennessee
  - Next Oncology, San Antonio, Texas
  - Next Virginia, Fairfax, Virginia
- Australia (3):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Peter MacCallum Cancer Centre, Parkville, Victoria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B Davis - Jewish General Hospital, Montreal, Quebec
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Centre Leon Berard, Lyon
  - Gustave Roussy, Villejuif
- Universitaetsklinikum Essen, Essen, Germany
- Italy (2):
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Centro Ricerche Cliniche Di Verona Societa responsabilita limitata, Verona
- Japan (3):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Fundacion Jimenez Diaz, Madrid, Spain
- Royal Marsden Hospital, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com